CLINICAL TRIAL: NCT02151045
Title: Comparison of a Cortivazol (ALTIM®) Infiltration of Posterior Epidural Space at L3-L4 Stage Versus an Epidural Infiltration of Cortivazol (ALTIM®) on Contact With Disco Radicular Conflict in Discal Sciatica - Controlled Randomized Trial With Double Blind Evaluation
Brief Title: Comparison of a Cortivazol (ALTIM®) Infiltration of Posterior Epidural Space at L3-L4 Stage Versus an Epidural Infiltration of Cortivazol (ALTIM®) on Contact With Disco Radicular Conflict in Discal Sciatica
Acronym: EPI-AMELIE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8708
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Discal Sciatica
Keywords: Epidural infiltration of Corticoids; L3-L4 stage; On contact of disco radicular conflict; Scan control

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non target epidural infiltration at L3-L4 stage (Active Comparator): In this control arm, there are patients with a non target posterior epidural space infiltration of corticoids done at L3-L4 stage on scan control.
  These patients must have a discal hernia confirmed by scanner or RMI
  Interventions: Procedure: Non target epidural infiltration done at L3-L4 stage
- Epidural infiltration on contact of disco radicular conflict (Experimental): In this experimental arm, there are patients with an epidural infiltration of corticoids done in lateral on contact of disco radicular conflict on scan control.
  These patients must have a discal hernia confirmed by scanner or RMI
  Interventions: Procedure: Epidural infiltration on contact of disco radicular conflict

INTERVENTIONS:
Procedure: Non target epidural infiltration done at L3-L4 stage — For patients included in control arm, a non target posterior epidural space infiltration of corticoids will be done at L3-L4 stage on scan control
  Arms: Non target epidural infiltration at L3-L4 stage
Procedure: Epidural infiltration on contact of disco radicular conflict — For patients included in experimental arm, an epidural infiltration of corticoids will be done in lateral on contact of disco radicular conflict on scan control.
  Arms: Epidural infiltration on contact of disco radicular conflict

SUMMARY:
In discal sciatica, after failure of medical treatment, the investigators propose frequently a spinal infiltration of corticoids the most closer of disco-radicular conflict. Recently, some cases of paraplegia during lumbar foraminal infiltrations have induce a reduction of indications of this type of infiltration. An alternative would be to propose a lateral epidural infiltration on contact with conflict.The objective of this study is to compare, in 112 patients with a less than 6 months discal sciatica, the efficacy on pain of a non target posterior epidural space infiltration of corticoids done at L3-L4 stage on scan control versus an epidural infiltration of the same corticoid done in lateral on contact of disco radicular conflict on scan control.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Aged from 18 to 65 years
* Affiliated or benefit from an insurance regimen
* Patient with a sciatic answering to the definition
* Discal sciatica more than 15 days and less than 6 months
* Discal hernia (scan or RMI)
* Negative BHCG and normal coagulation parameters

Exclusion Criteria:

* History of lumbar surgery
* Spinal infiltration of corticoids in 30 days before inclusion
* Iode allergy
* Anticoagulation therapy, unbalanced type 2 diabetes, instable HTA
* Motor loss < 4 (muscular testing)
* Sphincter disorder (cauda equida syndrome)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2012-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Pain evolution on analogic visual scale (EVA) ay Day 30 | at Day 30 after infiltration

SECONDARY OUTCOMES:
Pain evolution on analogic visual scal (EVA) at Day 7 | at day 7 after infiltration
Pain evolution on analogic visual scal (EVA) at month 3 | at month 3 after infiltration
Pain evolution on analogic visual scal (EVA) at month 6 | at month 6 after infiltration
Pain evolution on analogic visual scal (EVA) at month 12 | at month 12 after infiltration
drug consumption at day 7 | at day 7 after infiltration
drug consumption at month 3 | at month 3 after infiltration
drug consumption at month 6 | at month 6 after infiltration
drug consumption at month 12 | at month 12 after infiltration
functional handicap at Day 7 | at day 7 after infiltration
  functional handicap is assessed by auto-questionnary
functional handicap at month 3 | at month 3 after infiltration
  functional handicap is assessed by auto-questionnary
functional handicap at month 6 | at month 6 after infiltration
  functional handicap is assessed by auto-questionnary
functional handicap at month 12 | at month 12 after infiltration
  functional handicap is assessed by auto-questionnary
professional activity recovery at Day 7 | at day 7 after infiltration
  professional activity recovery is assessed by patient's interrogation: if recovery, conditions of recovery, date of recovery. If not recovery, for why?
professional activity recovery at month 3 | at month 3 after infiltration
  professional activity recovery is assessed by patient's interrogation: if recovery, conditions of recovery, date of recovery. If not recovery, for why?
professional activity recovery at month 6 | at month 6 after infiltration
  professional activity recovery is assessed by patient's interrogation: if recovery, conditions of recovery, date of recovery. If not recovery, for why?
professional activity recovery at month 12 | at month 12 after infiltration
  professional activity recovery is assessed by patient's interrogation: if recovery, conditions of recovery, date of recovery. If not recovery, for why?
new epidural infiltration or surgery of discal hernia at Day 7 | at day 7 after infiltration
new epidural infiltration or surgery of discal hernia at month 3 | at month 3 after infiltration
new epidural infiltration or surgery of discal hernia at month 6 | at month 6 after infiltration
new epidural infiltration or surgery of discal hernia at month 12 | at month 12 after infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Eric ET THOMAS, MD, Principal Investigator — CHU de Montpellier
Locations (2):
- France (2):
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU Carémeau, Nîmes